CLINICAL TRIAL: NCT07197658
Title: Prospective Healing Assessment After Application of Endodontic Microsurgery for Elimination of Apical Pathology By Use of Either a Rotary Bur for Osteotomy and Apical Root Resection, or Piezoelectric Unit for the Same Clinical Procedures
Brief Title: Healing After Endodontic Microsurgery Using a Rotary Bur Versus Piezoelectric Unit for Osteotomy and Root Resection
Acronym: BURVSPIEZO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Spyros Floratos, Principal Investigator, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 129586
Record Dates: First submitted 2025-08-24; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Periapical Periodontitis; Endodontic Microsurgery; Osteotomy
Keywords: Endodontic surgery; Piezosurgery; Bone window
MeSH Terms: conditions — Periapical Periodontitis | interventions — Piezosurgery

STUDY DESIGN:
Intervention Model Description: For this prospective investigation, patients will be randomly allocated into two groups. In the experimental group, endodontic microsurgery will be performed by use of a rotary bur for osteotomy and apical root resection.
  In the control group, piezoelectric surgery will be used for the same clinical procedures. All surgical procedures will be performed by one operator. Postsurgical healing as well as certain preoperative and postoperative parameters will be assessed and compared in the two groups. In a subgroup of patients having at least 2mm of intact buccal cortical bone thickness preoperatively, piezoelectric surgery will be used to prepare a rectangular buccal 'bone window'. The buccal bone thickness will be measured preoperatively on the coronal slices of the Cone Beam Computed Tomography (CBCT). After completing the root end filling, the bone window will be repositioned at the original position
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental Group) - Rotary bur (Experimental): Endodontic microsurgery will be performed by use of a rotary bur
  Interventions: Procedure: endodontic microsurgery / rotary bur osteotomy
- Group 2 (Control Group) - Piezoelectric unit (Active Comparator): Endodontic microsurgery will be performed by use of a piezoelectric unit
  Interventions: Procedure: Endodontic microsurgery / piezo osteotomy
- Bone Window subgroup (Active Comparator): 'Bone window' technique will be performed
  Interventions: Procedure: Endodontic microsurgery / bone window

INTERVENTIONS:
Procedure: endodontic microsurgery / rotary bur osteotomy — Endodontic microsurgery will be executed by use of a rotary bur
  Other Names: bur osteotomy; endodontic microsurgery
  Arms: Group 1 (Experimental Group) - Rotary bur
Procedure: Endodontic microsurgery / piezo osteotomy — Endodontic microsurgery will be performed by use of a piezosurgery unit
  Other Names: endodontic surgery; surgical endodontic retreatment; piezosurgery
  Arms: Group 2 (Control Group) - Piezoelectric unit
Procedure: Endodontic microsurgery / bone window — 'Bone window' technique will be performed by use of piezoelectric surgery
  Other Names: apical surgery; bone lid
  Arms: Bone Window subgroup

SUMMARY:
The goal of this clinical trial is to compare bone healing after using apical tooth microsurgery to remove root end infection, either by use of rotary burs for cutting bone and root end, or by use of piezoelectric surgery for the same procedures.

The main questions it aims to answer are:

* Is there a difference in bone healing and reformation between the two surgical procedures ?
* Is there a difference in bone healing between cutting the bone with a rotary bur and cutting the bone with the 'bone window' technique that uses piezoelectric unit ?

DETAILED DESCRIPTION:
The aim of this study is to prospectively compare postsurgical healing after the use of microsurgical technique to eliminate apical pathology, either by use of rotary burs for osteotomy and root resection, or by use of piezoelectric surgery for the same clinical procedures. Null hypothesis is that there is no difference in healing and buccal bone thickness reformation between the two surgical procedures Another purpose of the study is to prospectively evaluate healing after the application of a novel buccal bone preservation technique, called the 'bone window' technique. The technique will be applied in a subgroup of patients on maxillary and mandibular premolar and molar teeth with an intact buccal cortical bone and healing and buccal bone reformation will be assessed at follow up. Null hypothesis in this part, is that there is no difference in healing and buccal bone preservation between osteotomy with a bur and the 'bone window' technique.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older consenting to the surgical procedure as well as agreeing to preoperative, postoperative and at least one follow-up CBCT evaluation after 12 months
* Noncontributory medical history (American Society of Anesthesiologists class I and II)
* A history of previous endodontic treatment with radiographic presence of apical periodontitis
* A true endodontic lesion: microsurgical classification A, B, or C according to Kim and Kratchman, 2006.
* Lesion size 10 mm or smaller in diameter measured on preoperative CBCT
* Coronal restoration should be present at the time of follow up examination.

Exclusion Criteria:

* Nonconsenting patients and patients younger than 18 years of age
* Medical history with American Society of Anesthesiologists class III to V
* Insufficient coronal restoration
* Nonrestorability or traumatized teeth
* Teeth with microsurgical classification D, E, or F according to Kim and Kratchman, 2006.
* Mobility I or higher
* Radiographic presence of nonapical root resorption
* Teeth with a vertical root fracture or coronal/ midroot perforation
* Lesion size larger than 10 mm in diameter measured on preoperative CBCT
* Use of bone graft material for regeneration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Two dimensional radiographic bone healing | From execution of the microsurgical procedure to one year or later follow up examination
  Bone healing will be measured on periapical radiograph using well established two dimensional criteria for bone healing assessment. Molven's criteria categorize healing using periapical films into four categories: complete healing, incomplete healing, uncertain and unsatisfactory healing
Three dimensional radiographic bone healing | From execution of the microsurgical procedure to one year or later follow up examination
  Bone healing will be measured on Cone Beam Computed Tomography (CBCT) scan using well established three dimensional criteria for bone healing assessment. Penn 3D criteria categorize healing using CBCT scans into three categories: complete healing, limited and unsatisfactory healing

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Tsolakis, DMD,MS,PhD, Study Director — National Kapodistrian University of Athens
Locations (2):
- Greece (2):
  - Private Dental Office, Athens, Attica
  - Spyros Floratos Private Dental Office, Athens, Attica

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: IPD will be shared with researchers outside the study team after their request. Request has to be made to the study's principal investigator with explanation of the reason / scientific purpose the IPD is requested. IPD will be offered for conducting meta-analysis, systematic review studies on pertinent research study topics to the study conducted. Raw data with pseudonyms and numbering of participants, protocol data, results data, statistical analysis will be offered. The principal investigator of the study maintain all raw data in numbered folders with no information that reveals the participant identity. Numbered folders with no personal information of participants, tables , statistical analysis, anonymized excel files will be sent by email to other researchers after they sign a confidentiality statement for use of the data

REFERENCES:
- [Background] von Arx T, Janner SF, Hanni S, Bornstein MM. Agreement between 2D and 3D radiographic outcome assessment one year after periapical surgery. Int Endod J. 2016 Oct;49(10):915-25. doi: 10.1111/iej.12548. Epub 2015 Oct 8. PMID 26356580
- [Background] Chen I, Karabucak B, Wang C, Wang HG, Koyama E, Kohli MR, Nah HD, Kim S. Healing after root-end microsurgery by using mineral trioxide aggregate and a new calcium silicate-based bioceramic material as root-end filling materials in dogs. J Endod. 2015 Mar;41(3):389-99. doi: 10.1016/j.joen.2014.11.005. Epub 2015 Jan 14. PMID 25596728
- [Background] Hirsch V, Kohli MR, Kim S. Apicoectomy of maxillary anterior teeth through a piezoelectric bony-window osteotomy: two case reports introducing a new technique to preserve cortical bone. Restor Dent Endod. 2016 Nov;41(4):310-315. doi: 10.5395/rde.2016.41.4.310. Epub 2016 Jul 5. PMID 27847753
- [Background] Khoury F, Hensher R. The bony lid approach for the apical root resection of lower molars. Int J Oral Maxillofac Surg. 1987 Apr;16(2):166-70. doi: 10.1016/s0901-5027(87)80125-x. PMID 3110314
- [Background] Vercellotti T, De Paoli S, Nevins M. The piezoelectric bony window osteotomy and sinus membrane elevation: introduction of a new technique for simplification of the sinus augmentation procedure. Int J Periodontics Restorative Dent. 2001 Dec;21(6):561-7. PMID 11794567
- [Background] Yaman Z, Suer BT. Piezoelectric surgery in oral and maxillofacial surgery. Annals of Oral and Maxillofacial Surgery. 2013; 1:1-9
- [Background] Chopra P, Chopra P. Piezosurgery and its applications in Periodontology and Implantology. International Journal of Contemporary Dentistry. 2011;2(4): 16-24
- [Background] Rashad A, Kaiser A, Prochnow N, Schmitz I, Hoffmann E, Maurer P. Heat production during different ultrasonic and conventional osteotomy preparations for dental implants. Clin Oral Implants Res. 2011 Dec;22(12):1361-5. doi: 10.1111/j.1600-0501.2010.02126.x. Epub 2011 Mar 21. PMID 21435005
- [Background] Song M, Kim E. A prospective randomized controlled study of mineral trioxide aggregate and super ethoxy-benzoic acid as root-end filling materials in endodontic microsurgery. J Endod. 2012 Jul;38(7):875-9. doi: 10.1016/j.joen.2012.04.008. Epub 2012 May 16. PMID 22703646
- [Background] Tsesis I, Rosen E, Schwartz-Arad D, Fuss Z. Retrospective evaluation of surgical endodontic treatment: traditional versus modern technique. J Endod. 2006 May;32(5):412-6. doi: 10.1016/j.joen.2005.10.051. PMID 16631838
- [Background] Setzer FC, Shah SB, Kohli MR, Karabucak B, Kim S. Outcome of endodontic surgery: a meta-analysis of the literature--part 1: Comparison of traditional root-end surgery and endodontic microsurgery. J Endod. 2010 Nov;36(11):1757-65. doi: 10.1016/j.joen.2010.08.007. Epub 2010 Sep 17. PMID 20951283
- [Background] Safi C, Kohli MR, Kratchman SI, Setzer FC, Karabucak B. Outcome of Endodontic Microsurgery Using Mineral Trioxide Aggregate or Root Repair Material as Root-end Filling Material: A Randomized Controlled Trial with Cone-beam Computed Tomographic Evaluation. J Endod. 2019 Jul;45(7):831-839. doi: 10.1016/j.joen.2019.03.014. Epub 2019 May 9. PMID 31078325
- [Background] Floratos S, Kim S. Modern Endodontic Microsurgery Concepts: A Clinical Update. Dent Clin North Am. 2017 Jan;61(1):81-91. doi: 10.1016/j.cden.2016.08.007. PMID 27912820
- [Background] Kim S, Kratchman S. Modern endodontic surgery concepts and practice: a review. J Endod. 2006 Jul;32(7):601-23. doi: 10.1016/j.joen.2005.12.010. Epub 2006 May 6. PMID 16793466

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT07197658/Prot_SAP_000.pdf